CLINICAL TRIAL: NCT03410394
Title: Registre Tumeurs Endocrine - Eurocrine
Brief Title: Registry of Endocrine Tumors (Thyroid, Parathyroid, Adrenal, Endocrine Pancreas, Endocrine Digestive Tube)
Acronym: eurocrine
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laurent BRUNAUD, investigator, Central Hospital, Nancy, France
Other Study IDs: N° CCTIRS :15.291 Version N°3
Record Dates: First submitted 2018-01-10; First posted 2018-01-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Endocrine Tumor
Keywords: adrenal; thyroid; parathyroid; endocrine pancreas; endocrine digestive tube
MeSH Terms: conditions — Endocrine Gland Neoplasms; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — samples from tumor specimen. All patients signed a specific and validated form allowing the collection of samples with DNA (CNIL N° DC2014-2114)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- registry of endocrine tumors: * Patients who undergo thyroid surgical procedures. This registry was declared at the commission national informatique et libertés (CNIL) with the number R2015-22.
  * Patients who undergo parathyroid surgical procedures. This registry was declared at the commission national informatique et libertés (CNIL) with the number R2015-23
  * Patients who undergo adrenal surgical procedures. This registry was declared at the commission national informatique et libertés (CNIL) with the number R2015-24
  * Patients who undergo pancreatic and digestive surgical procedures. This registry was declared at the commission national informatique et libertés (CNIL) with the number R2015-26

SUMMARY:
This registry aims to collect informations about patients with endocrine tumors (Thyroid, Parathyroid, Adrenal, Endocrine Pancreas, Endocrine Digestive Tube) who undergo endocrine surgical procedures. This registry is part of the Eurocrine Project.

DETAILED DESCRIPTION:
The EUROCRINE project aims to decrease morbidity and mortality of rare endocrine tumours, by means of a pan-European database. Recording and accessing data at the European level, makes it possible to identify these tumours, which cannot be distinguished at local or national level, because of their extreme rarity. Dissemination of results aims to raise clinical standards and reduce differences in practise between clinics and member states, and thereby diminish morbidity and mortality. Comparison of practice and outcomes will be especially interesting for centres wanting to improve their standards to what is currently considered best practice. EUROCRINE will be a key means by which the medical profession, researchers, health policy makers, and not least patients, can benefit from an increase in knowledge related to diagnosis, treatment, and future clinical research in the field of rare endocrine tumours.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo surgical procedures for endocrine tumors at the University Nancy Brabois Hospital

Exclusion Criteria:

* unable to receive clear information
* refusal to sign the consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who undergo surgical procedures for endocrine tumors at CHU Nancy Brabois (University hospital)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications (endocrine surgical procedure) | 12 months after surgical procedure
  morbidity rate in percentage (%)

SECONDARY OUTCOMES:
Postoperative complications severity (endocrine surgical procedure) | 12 months after surgical procedure
  Dindo-Clavien classification in percentage (%)
Postoperative mortality (endocrine surgical procedure) | 12 months after surgical procedure
  mortality rate in percentage (%)
CT imaging before endocrine surgical procedure (Tumor characteristics) | Baseline
  Density in Hounsfield unit (HU)
CT imaging before endocrine surgical procedure (Coronary artery score) | Baseline
  CAC score in Agatston score unit (HU)
CT imaging before endocrine surgical procedure (Sarcopenia) | preoperative period
  Evaluation of sarcopenia using L3 skeletal muscle index (in cm²/m²)
Bone mineral density | Baseline
  dual-energy x-ray absorptiometry (DEXA) (in T-score unit)
Intraoperative systolic arterial pressure | Intraoperative
  systolic arterial pressure (in mmHg)
Intraoperative diastolic arterial pressure | Intraoperative
  diastolic arterial pressure (in mmHg)
Parathormone plasma levels | Baseline and up to 12 months after surgical procedure
  Parathormone (in pg/mL)
Aldosterone plasma levels | Baseline and up to 12 months after surgical procedure
  Aldosterone (in pmol/L)
Plasma renin activity | Baseline and up to 12 months after surgical procedure
  Renin (in μIU/mL)
Plasma free metanephrines | Baseline and up to 12 months after surgical procedure
  metanephrines (in nmol/L)
PET scanning | Baseline
  standardized uptake values (SUV tumor / SUV liver ratio)

CONTACTS AND LOCATIONS:
Overall Officials: laurent Brunaud, Principal Investigator — University of Lorraine
Locations (1):
- CHU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greilsamer T, Nomine-Criqui C, Thy M, Ullmann T, Zarnegar R, Bresler L, Brunaud L. Robotic-assisted unilateral adrenalectomy: risk factors for perioperative complications in 303 consecutive patients. Surg Endosc. 2019 Mar;33(3):802-810. doi: 10.1007/s00464-018-6346-2. Epub 2018 Jul 11. PMID 29998394
- See also: EUROCRINE WEB SITE — https://eurocrine.eu/